CLINICAL TRIAL: NCT05939947
Title: A Double-Blind Placebo-Controlled Randomised Phase 1b Study of the Pharmacokinetics of ALE.F02 in Patients With Advanced Liver Fibrosis and/or With Mild Cirrhosis
Brief Title: A Clinical Trial of ALE.F02 in Patients With Advanced Liver Fibrosis and/or With Mild Cirrhosis
Acronym: FEGATO-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alentis Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: ALE.F02.02
Record Dates: First submitted 2023-06-21; First posted 2023-07-11 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Advanced Liver Fibrosis; Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: Thirty-eight patients will receive 3 doses of ALE.F02 or matching placebo, administered once every second week as a continuous intravenous (IV) infusion to a total of 3 doses per patient at the same dose level. The 4 cohorts are enrolled in a staggered sequence and escalated upon review and approval of a Safety Review Committee: Cohort 1 (low dose) (4:2 active:placebo), Cohort 2 (intermediate dose) (8:4), Cohort 3 (intermediate dose) (8:2), Cohort 4 (high dose) (8:2).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALE.F02 (Experimental): Patients will receive 3 doses of ALE.F02 administered once every second week as a continuous intravenous (IV) infusion to a total of 3 doses.
  Interventions: Drug: ALE.F02
- Placebo (Placebo Comparator): Patients will receive 3 doses of matching placebo administered once every second week as a continuous intravenous (IV) infusion to a total of 3 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALE.F02 — Continuous intravenous (IV) infusion administered once every second week to a total of 3 doses.
  Arms: ALE.F02
Drug: Placebo — Continuous intravenous (IV) infusion administered once every second week to a total of 3 doses.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate how a human body processes ALE.F02 (pharmacokinetics profile) in patients with impaired liver function.

ELIGIBILITY:
Principal Inclusion Criteria:

* Outpatients between 18 and 80 years
* Have been diagnosed with advanced liver fibrosis or mild cirrhosis attributable to NASH, ALD, or following a sustained virological response to treatment for hepatitis C
* Have an ELF Score of at least 9.5 but no more than 13
* Have stable hepatic impairment, defined as no clinically significant change in disease status, and no previous liver cirrhosis decompensation episodes
* Body weight within the range of 50.0 kg to 140.0 kg
* Clinical frailty score <6

Principal Exclusion Criteria:

* Child-Pugh score ≥7, as determined at screening
* MELD score ≥12, as determined at screening
* Estimated glomerular filtration rate <60 mL/min per the CKD-EPI creatinine-cystatin C equation
* Current or history of HCC
* Be suffering from or have symptoms of an acute or chronic infection
* Have active hepatitis C infection
* Other causes of liver disease including, but not limited to, hepatitis B, autoimmune disorders drug-induced hepatotoxicity, Wilson's disease, iron overload, and alpha-1-antitryspin deficiency, based on medical history review.
* Is a woman of childbearing potential

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) profile of ALE.F02 in patients with advanced liver fibrosis and/or with mild cirrhosis using noncompartmental analysis. | Baseline to Day 14 and Day 29 to Day 72
  Maximum Serum Concentration [Cmax]
Pharmacokinetics (PK) profile of ALE.F02 in patients with advanced liver fibrosis and/or with mild cirrhosis using noncompartmental analysis. | Baseline to Day 14 and Day 29 to Day 72
  Time of Maximum Serum Concentration [Tmax]
Pharmacokinetics (PK) profile of ALE.F02 in patients with advanced liver fibrosis and/or with mild cirrhosis using noncompartmental analysis. | Baseline to Day 14 and Day 29 to Day 72
  Area under the serum concentration versus time curve [AUC0-tau, AUC0-inf]

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events of ALE.F02 in patients with advanced liver fibrosis and/or with mild cirrhosis. | Baseline to Day 72
  Incidence of Treatment-Emergent Adverse Events assessed by CTCAE v5.0 criteria
  Incidence of Serious Adverse Events assessed by CTCAE v5.0 criteria
Pharmacodynamic (PD) profile of ALE.F02 in patients with advanced liver fibrosis and/or with mild cirrhosis. | Baseline to Day 72
  Relative change (%) of serum levels of PRO-C3 between baseline and the EOT.
  Relative change (%) of serum levels of tissue inhibitor of matrix metalloproteinase [TIMP1] between baseline and the EOT.
  Relative change (%) of serum levels of hyaluronic acid between baseline and the EOT.
  Relative change (%) of serum levels of procollagen III amino-terminal peptide [PIIINP] between baseline and the EOT.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Manenti, MD, Study Director — Alentis Therapeutics AG
Locations (6):
- American Research Corporation, San Antonio, Texas, United States
- APEX GmbH, Munich, Germany
- Romania (2):
  - ARENSIA Exploratory Medicine S.R.L., Bucharest
  - ARENSIA Exploratory Medicine S.R.L. - Cluj-Napoca, Cluj-Napoca
- Slovakia (2):
  - Summit Clinical Research, Bratislava
  - Summit Clinical Research, Malacky

IPD SHARING:
Plan to Share IPD: No